CLINICAL TRIAL: NCT03736330
Title: A Study of Anti-PD-1( Pembrolizumab) Combinations of D-CIK (Cytokine-induced Killer Cells Are Stimulated Using Mature Dendritic Cells) Immunotherapy and Axitinib in Advanced Ranal Carcinoma
Brief Title: A Study of Anti-PD-1 Combinations of D-CIK Immunotherapy and Axitinib in Advanced Ranal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Director Of Urology, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-FXY-023-Urology
Record Dates: First submitted 2018-11-01; First posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Renal Cancer Metastatic
Keywords: Ranal Carcinoma; Immunotherapy; Axitinib

STUDY DESIGN:
Intervention Model Description: Autologous D-CIK (1.0-1.5*10^10 cells) will be transferred to patients via intravenous infusion. Before cell transfer, D-CIK were incubated with anti-PD-1 antibody.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combinations treatment (Experimental): Drug: Axitinib 5mg orally twice a day Combination Treatment：Anti-PD-1 Combinations of D-CIK Immunotherapy
  Interventions: Biological: Combinations treatment

INTERVENTIONS:
Biological: Combinations treatment — Autologous dendritic and cytokine-induced killer cells (D-CIK)(1.0-1.5*10^10 cells)were incubated with low dose anti-PD-1 antibody（pembrolizumab, Merck & Co., Inc.） and were transferred to participants via intravenous infusion .
  Other Names: pembrolizumab(Merck & Co., Inc.)

SUMMARY:
Phase II clinical trial to investigate the safety, clinical activity and toxicity of combinations of D-CIK and low dose anti-PD-1 antibody in patients with metastatic renal cell carcinoma treated with axitinib.

DETAILED DESCRIPTION:
This is a phase II, single arm study to investigate the safety and efficacy of pembrolizumab-activated autologous D-CIK cells (CIK:Cytokine-induced killer, D-CIK:CIK cells are stimulated using mature dendritic cells) with Axitinib in patients with advanced kidney cancer.

Heparinized peripheral blood was obtained from participants over a 1-week period. PBMCs(Peripheral blood mononuclear cells) were separated by Ficoll-Hypaque gradient centrifugation, suspended in X-VIVO 15 serum-free medium, and culture with 1000 U/ml rhIFN-γfor the first 24 h, followed by stimulation with 100 ng/ml OKT-3 , 1000 U/ml rhIL-2 and 100 U/ml IL-1α to activate the CIK.Dendritic cells were incubated with CIK. Fresh medium containing 1000 U/ml rhIL-2 was added every 2 days and the cell density was maintained at 2×10^6 cells/mL.D-CIK were harvested, washed, and resuspended after culture for 14 days. Before cell transfer,D-CIK were incubated with anti-PD-1 antibody(Pembrolizumab (Merck & Co., Inc.) is a humanized IgG4 anti-PD-1 monoclonal antibody that binds to PD-1 to prevent it from engaging with PD-L1 or PD-L2.), and a fraction of the D-CIK were collected to assess their number, phenotype, and viability of cells, and to test for possible contamination by bacteria, fungi, or endotoxins. Then, autologous D-CIK (1.0-1.5*10^10 cells) were transferred to patients via intravenous infusion.

The present study was designed with Simon's best two stage study to explore the efficacy and safety of low-dose pembrolizumab in the treatment of patients with advanced renal cancer by D-CIK re-transfusion combined with Axitinib in vitro. The expected effective rate of the combined treatment is set at 60%, and if the effective rate is less than 30%, the effective rate of the combined treatment is considered to be at an undesirable level. The best two-stage design is 3/8, 10/24. In the first stage, 8 patients need to be treated. If the number of effective cases is less than 3, the combined treatment is deemed ineffective and the trial needs to be terminated. If the number of effective cases is more than 3, the phase II trial will be continued, and a total of 24 subjects need to be included.

ELIGIBILITY:
Inclusion Criteria:

* advanced renal clear cell carcinoma confirmed by pathology: high-volume disease without systemic treatment(including primary lesion unable to surgery, multiple lymph node metastases or distant metastases), or achieved disease progression after treatment by the anti-angiogenesis therapy (TKI or mTOR inhibitors) or by cytokines or combination therapy
* Predicted survival >=3 months
* At least 1 measurable lesion

High-volume disease（meet one of the following criteria）:1. More than 3 sites of lesions with or without primary lesions, and at least 1 lesion routine CT or spiral CT scan >=3cm; 2. Unresected primary lesions (> 10cm), accompanied by 2 metastatic lesions; 3. After nephrectomy, single metastasis, at least 3 metastases, and at least one lesion > 2cm; 4. After nephrectomy, multiple metastatic(>3 organs) and at least one lesion > 2cm.

Exclusion Criteria:

* Prior treatment with anti-PD-1/PD-L1/PD-L2 antibody and Axitinib
* Hypersensitivity to recombinant humanized anti-PD-1 monoclonal Abm or its components
* Severe cardiovascular and cerebrovascular diseases, uncontrollable severe hypertension and diabetes, severe renal insufficiency or uremia
* Long-term use of immunosuppressive agents after organ transplantation
* Immunosuppressive drugs are currently in use
* People with a clear and serious infection
* Predicted survival<3 months
* Patients with T cell lymphoma, myeloma
* Patients with autoimmune diseases
* HIV positive, or other immunodeficiency diseases
* Pregnant or nursing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-09-08 (Actual); Primary Completion 2020-10-08 (Estimated); Study Completion 2021-11-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR）by irRC and RECIST 1.1 | 3 years
  The treatment effect of Anti-PD-1 combinations of D-CIK immunotherapy and axitinib,will be assessed using irRC and RECIST 1.1 to determine tumor response.

SECONDARY OUTCOMES:
Progression-free Survival（PFS）by irRC and RECIST 1.1 | 3 years
  The treatment effect of Anti-PD-1 combinations of D-CIK immunotherapy and axitinib, will be assessed using irRC and RECIST 1.1 to determine progression-free survival time.
Overall Survival (OS) by irRC and RECIST 1.1 | 3 years
  The treatment effect of Anti-PD-1 combinations of D-CIK immunotherapy and axitinib, will be assessed using irRC and RECIST 1.1 to determine overall survival time.
Duration of Response (DOR) by irRC and RECIST 1.1 | 3 years
  The treatment effect of Anti-PD-1 combinations of D-CIK immunotherapy and axitinib, will be assessed using irRC and RECIST 1.1 to determine duration of response.
The quality of life by EQ-5D-5L and NCCN-FACT FKSI-19 v2.0. | 3 years
  The treatment effect of Anti-PD-1 combinations of D-CIK immunotherapy and axitinib, will be assessed using EQ-5D-5L and NCCN-FACT FKSI-19 v2.0.to determine the quality of life.
Severity of adverse events as assessed by CTCAE v4.0 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Fangjian Zhou, MD.PhD, Principal Investigator — Director of Urology,Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
We did not decide whether to share the subject's personal information

REFERENCES:
- [Result] Rini BI, Escudier B, Tomczak P, Kaprin A, Szczylik C, Hutson TE, Michaelson MD, Gorbunova VA, Gore ME, Rusakov IG, Negrier S, Ou YC, Castellano D, Lim HY, Uemura H, Tarazi J, Cella D, Chen C, Rosbrook B, Kim S, Motzer RJ. Comparative effectiveness of axitinib versus sorafenib in advanced renal cell carcinoma (AXIS): a randomised phase 3 trial. Lancet. 2011 Dec 3;378(9807):1931-9. doi: 10.1016/S0140-6736(11)61613-9. Epub 2011 Nov 4. PMID 22056247
- [Result] Du Four S, Maenhout SK, De Pierre K, Renmans D, Niclou SP, Thielemans K, Neyns B, Aerts JL. Axitinib increases the infiltration of immune cells and reduces the suppressive capacity of monocytic MDSCs in an intracranial mouse melanoma model. Oncoimmunology. 2015 Jan 22;4(4):e998107. doi: 10.1080/2162402X.2014.998107. eCollection 2015 Apr. PMID 26137411
- [Result] Mahoney KM, Rennert PD, Freeman GJ. Combination cancer immunotherapy and new immunomodulatory targets. Nat Rev Drug Discov. 2015 Aug;14(8):561-84. doi: 10.1038/nrd4591. PMID 26228759
- [Result] Lee JH, Lee JH, Lim YS, Yeon JE, Song TJ, Yu SJ, Gwak GY, Kim KM, Kim YJ, Lee JW, Yoon JH. Adjuvant immunotherapy with autologous cytokine-induced killer cells for hepatocellular carcinoma. Gastroenterology. 2015 Jun;148(7):1383-91.e6. doi: 10.1053/j.gastro.2015.02.055. Epub 2015 Mar 4. PMID 25747273
- [Result] Chen CL, Pan QZ, Weng DS, Xie CM, Zhao JJ, Chen MS, Peng RQ, Li DD, Wang Y, Tang Y, Wang QJ, Zhang ZL, Zhang XF, Jiang LJ, Zhou ZQ, Zhu Q, He J, Liu Y, Zhou FJ, Xia JC. Safety and activity of PD-1 blockade-activated DC-CIK cells in patients with advanced solid tumors. Oncoimmunology. 2018 Jan 10;7(4):e1417721. doi: 10.1080/2162402X.2017.1417721. eCollection 2018. PMID 29632736